CLINICAL TRIAL: NCT03769896
Title: Nabilone for Non-motor Symptoms in Parkinson's Disease: A Randomized Placebo-controlled, Double-blind, Parallel-group, Enriched Enrolment Randomized Withdrawal Study
Brief Title: Nabilone for Non-motor Symptoms in Parkinson's Disease
Acronym: NMS-Nab
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Principal Investigator, Klaus Seppi, MD, Principal Investigator, Medical University Innsbruck
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1.4
Record Dates: First submitted 2018-12-06; First posted 2018-12-10 (Actual); Results first posted 2021-03-02 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-02

CONDITIONS: Parkinson Disease
Keywords: Parkinson´s Disease; cannabinoids; non-motor symptoms
MeSH Terms: conditions — Parkinson Disease | interventions — nabilone

STUDY DESIGN:
Intervention Model Description: randomized placebo-controlled, double-blind, parallel-group, enriched enrolment randomized withdrawal study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: placebo-controlled, double-blind, parallel-group with 1 : 1 randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Active Comparator): Nabilone 0.25 mg
  Interventions: Drug: Nabilone 0.25 mg
- Placebo Group (Placebo Comparator): Placebo (corn starch)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nabilone 0.25 mg — capsules, 0.25 mg up to 2 mg of nabilone taken orally on a daily basis
  Arms: Treatment Group
Drug: Placebo — capsule, corn starch, daily basis
  Arms: Placebo Group

SUMMARY:
This is a randomized placebo-controlled, double-blind, parallel-group, enriched enrollment randomized withdrawal study assessing the efficacy and safety of nabilone for non-motor symptoms in patients with Parkinson´s Disease. Nabilone is an analogue of tetrahydrocannabinol (THC), the psychoactive component of cannabis. Nabilone acts as a partial agonist on both Cannabinoid 1 (CB1) and Cannabinoid 2 (CB2) receptor in humans and therefore mimics the effect of THC but with more predictable side effects and less euphoria.

Part 1 is an open-label dose adjustment phase of the study. In eligible patients, a screening period is followed by an open-label nabilone dose optimization phase and a stable phase for at least 1 week. Treatment responders will be included in Part 2 of the study (randomized placebo-controlled, double-blind, parallel-grouped).

Part 2 is the placebo-controlled, double-blind, parallel-group randomized withdrawal phase of the study.

DETAILED DESCRIPTION:
This is a randomized placebo-controlled, double-blind, parallel-group, enriched enrollment randomized withdrawal study assessing the efficacy and safety of nabilone for non-motor symptoms in patients with Parkinson´s Disease. Nabilone is an analogue of tetrahydrocannabinol (THC), the psychoactive component of cannabis. Nabilone acts as a partial agonist on both Cannabinoid 1 (CB1) and Cannabinoid 2 (CB2) receptor in humans and therefore mimics the effect of THC but with more predictable side effects and less euphoria.

Part 1 is the open-label dose adjustment phase of the study. In Part 1, eligible subjects, who have signed the informed consent form at the screening visit, will receive open-label nabilone starting with a dosage of 0.25 mg in the evening. During dose titration and optimization, nabilone will be titrated in 0.25 mg increments (increase by 0.25 mg/ every one to four days) up to a maximum dose of 1 mg twice daily. Patients should be on a stable nabilone dose for at least 1 week afterwards until Baseline Visit (V 0).

Part 2 is the placebo-controlled, double-blind, parallel-group randomized withdrawal phase of the study. At Baseline Visit, treatment responders will be included in Part 2 of the study (randomized placebo-controlled, double-blind, parallel-grouped). Responders are randomized in a 1:1 ratio at Baseline Visit to receive either nabilone or matching placebo for 4 weeks + 2 days. The placebo-controlled, double-blind, randomized withdrawal phase will end with a clinic visit (Termination Visit V 1). Following this, the study medication will be tapered in all patients. During this period the patients will receive phone calls every other day. A Safety Telephone Call and a Safety Follow-Up Visit will be performed.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible for the study subjects must meet all inclusion criteria:

1. Age ≥30 years
2. Diagnosis of Parkinson´s Disease (PD): PD should be either de novo or on stable medication without disturbing motor fluctuations or dyskinesia.
3. NMS with a score of ≥4 on MDS-UPDRS Part 1. One of the following domains have to be affected with a score ≥2: 1.4 (anxious mood) or 1.9 (pain)
4. On a stable regimen of anti-parkinson medications for at least 30 days prior to screening and willing to continue the same doses and regimens during study participation
5. Any other current and allowed prescription/non-prescription medications and/or nutritional supplements taken regularly must have been at a stable dose and regimen for at least 30 days prior to screening, and subject must be willing to continue the same doses and regimens during study participation
6. Patient is informed and had enough time and opportunity to think about his/her participation in the study and has signed a current Institutional Review Board-approved informed consent form
7. Contraception

   1. Women of childbearing potential must use or attest an acceptable method* of contraception starting 4 weeks prior to study drug administration and for a minimum of 1 month after study completion.
   2. Men with a potentially fertile partner must be willing to use an acceptable method of contraception for the duration of the study and for 3 months after study drug discontinuation or have had a vasectomy.

Exclusion Criteria:

Patients with any of the following characteristics will be excluded from entering the study:

1. Patient previously participated in any study with nabilone.
2. Current use of cannabinoids or use of cannabinoids within 30 days prior to screening.
3. Patient is currently participating in or has participated in another study of investigational products within 30 days prior to screening.
4. Patient has any form of secondary or atypical parkinsonism (e.g., drug-induced, post stroke).
5. Patient presents with motor complications which are, based on the investigator's judgment, not adequately controlled (i.e. a score ≥2 on one of the items of the MDS-UPDRS Part IV at screening)
6. Hoehn and Yahr stage > 3
7. Evidence of disturbing (i.e. requiring treatment) impulse control disorder in the participant. Can be resolved through a structural interview during screening period.
8. History of neurosurgical intervention for PD
9. presence of symptomatic orthostatic hypotension at screening (MDS-UPDRS 1.12 > 2)
10. Use of prohibited medication (e.g. benzodiazepines (except for clonazepam up to a maximum of 1.5 mg per d), lithium, opioids, buspirone, muscle relaxing agents, central nervous system depressing substances, ...)
11. Patients with laboratory values that are out-of-range at Screening (or within 4 weeks prior to Screening) and haven´t been reviewed and documented as not clinically significant by the investigator. Lab Tests can be repeated for confirmation.
12. Patients with known or newly diagnosed sinus tachycardia in ECG evaluation at Screening or within 4 weeks prior to Screening.
13. presence of an acute or chronic major psychiatric disorder (e.g., Major Depressive Disorder, psychosis) or symptom (e.g., hallucinations, agitation, paranoia) (MDS-UPDRS 1.2 and/or 1.3 > 2)
14. Patients who had a recent suicidal attempt (active, interrupted, aborted) within the past five years or report suicidal ideation within the past 6 months.
15. presence of dementia (MDS-UPDRS 1.1 > 2, Mini-Mental State Examination of <24 at the Screening visit)
16. clinically significant or unstable medical or surgical condition at Screening or Baseline visit that may preclude safety and the completion of the study participation (based on the investigator's judgment).
17. Patients with moderate or severe hepatic or renal impairment.
18. Patient has a history of chronic alcohol or drug abuse within the last 2 years.
19. women of child-bearing potential who do not practice an acceptable method of birth control
20. Pregnant women or women planning to become pregnant during the course of the study and nursing women.
21. Patients who are knowingly hypersensitive to any of the components of the investigational medicinal product or excipients.
22. Patient is legally incapacitated or persons held in an institution by legal or official order
23. Persons with any kind of dependency on the investigator or employed by the Sponsor or investigator

Ages: 30 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2017-10-03 (Actual); Primary Completion 2019-07-15 (Actual); Study Completion 2019-07-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurology - Medical University Innsbruck, Innsbruck, Tyrol, Austria

IPD SHARING:
Plan to Share IPD: No
The results of this study will be published according to the principles of publication policy. There are no arrangements on publication issues with subsiding parties.

REFERENCES:
- [Derived] Peball M, Seppi K, Krismer F, Knaus HG, Spielberger S, Heim B, Ellmerer P, Werkmann M, Poewe W, Djamshidian A. Effects of Nabilone on Sleep Outcomes in Patients with Parkinson's Disease: A Post-hoc Analysis of NMS-Nab Study. Mov Disord Clin Pract. 2022 May 31;9(6):751-758. doi: 10.1002/mdc3.13471. eCollection 2022 Aug. PMID 35937495
- [Derived] Peball M, Krismer F, Knaus HG, Djamshidian A, Werkmann M, Carbone F, Ellmerer P, Heim B, Marini K, Valent D, Goebel G, Ulmer H, Stockner H, Wenning GK, Stolz R, Krejcy K, Poewe W, Seppi K; Collaborators of the Parkinson's Disease Working Group Innsbruck. Non-Motor Symptoms in Parkinson's Disease are Reduced by Nabilone. Ann Neurol. 2020 Oct;88(4):712-722. doi: 10.1002/ana.25864. Epub 2020 Aug 31. PMID 32757413

RESULTS

PARTICIPANT FLOW:
Recruitment Details: location: Medical Clinic, period: October 2017 to July 2019
Pre-assignment Details: Phase 1: open-label nabilone titration (0.25mg - 2mg). Phase 2: double-blind phase There was one screening failure due to the use of prohibited concomitant medication.
Period: Open-label Phase
Arm/Group | Treatment Group | Placebo Group
Started | 47 | 0
Completed | 38 | 0
Not Completed | 9 | 0
Not completed — Lack of Efficacy | 5 | 0
Not completed — Adverse Event | 3 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Double-blind Treatment Phase
Arm/Group | Treatment Group | Placebo Group
Started (refers to the double-blind treatment phase) | 19 | 19
Completed (refers to the double-blind treatment phase) | 19 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: baseline characteristics (as assessed at the screening visit) for the 38 randomized patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Group | Placebo Group | Total
Number analyzed (Participants) | 19 | 19 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.38 (7.94) | 63.95 (8.04) | 65.05 (8.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 5 | 14
  Male | 10 | 14 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 19 | 19 | 38
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 00 | 0
  White | 19 | 19 | 38
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Austria | 19 | 19 | 38
Disease duration [Mean (Standard Deviation); unit: years] | 7.83 (5.47) | 7.39 (5.14) | 7.61 (5.24)
Hoehn and Yahr Scale [Mean (Standard Deviation); unit: units on a scale] — Hoehn and Yahr scale:
  * is used to assess the severity / disease stage of Parkinson´s disease patients
  * 5-point Likert scale
  * the total score ranges from a minimum of 0 to a maximum of 5
  * higher values indicate worse status
  * The total score values are reported in this table.
  units on a scale | 1.84 (0.50) | 1.95 (0.41) | 1.89 (0.45)
MDS-UPDRS Total Score [Mean (Standard Deviation); unit: units on a scale] — Movement Disorders Society - Unified Parkinson´s Disease Rating Scale (MDS-UPDRS)
  * Total score reported is the sum of Parts I to IV.
  * Part I minimum points: 0, maximum points: 52, Part II: minimum points: 0, maximum points: 52, Part III: minimum points: 0, maximum points: 132, Part IV: minimum points: 0, maximum points: 24.
  * Total MDS-UPDRS score: minimum: 0, maximum: 260.
  * Higher score values indicate a worse outcome.
  units on a scale | 52.05 (22.97) | 52.05 (14.75) | 52.05 (19.04)
MDS-UPDRS-I [Mean (Standard Deviation); unit: units on a scale] — Movement Disorders Society - Unified Parkinson´s Disease Rating Scale (MDS-UPDRS) Part I
  * minimum points: 0, maximum points: 52.
  * higher score values indicate a worse outcome.
  units on a scale | 13.53 (4.39) | 12.26 (5.85) | 12.89 (5.14)

OUTCOME MEASURES:

1. Primary Outcome: Changes of Non-motor Symptoms
Description: Changes in Movement Disorders Society - Unified Parkinson´s Disease Rating Scale (MDS-UPDRS) Part I minimum points: 0, maximum points: 52, higher score values indicate a worse outcome.
Time Frame: from baseline to 4 weeks + 2 days
Measure: Mean (90% Confidence Interval); unit: units on a scale
Arm/Group | Treatment Group | Placebo Group
Number analyzed (Participants) | 19 | 19
units on a scale | 1.00 [-0.16 to 2.16] | 2.63 [1.53 to 3.74]

2. Secondary Outcome: Changes in Motor and Different Non-motor Symptoms of PD
Description: Changes in Movement Disorders Society - Unified Parkinson´s Disease Rating Scale (MDS-UPDRS) Part II: minimum points: 0, maximum points: 52, higher score values indicate a worse outcome.
  Part III: minimum points: 0, maximum points: 132, higher score values indicate a worse outcome.
Time Frame: from baseline to 4 weeks + 2 days
Measure: Mean (90% Confidence Interval); unit: units on a scale
Arm/Group | Treatment Group | Placebo Group
Number analyzed (Participants) | 19 | 19
units on a scale
  MDS-UPDRS II | 0.47 [-0.37 to 1.31] | 0.90 [-0.35 to 2.14]
  MDS-UPDRS III | 0.53 [-2.24 to 3.29] | 2.63 [0.25 to 5.02]

3. Secondary Outcome: Changes in Different Domains of Non-motor Symptoms of PD
Description: mood/anxiety domain of MDS-UPDRS Part I (items 1.3 and 1.4) and different other domains of NMSS and MDS-UPDRS part I Each items scores 0 to 4 points with higher score values indicating a worse outcome.
Time Frame: from baseline to 4 weeks + 2 days
Measure: Mean (90% Confidence Interval); unit: units on a scale
Arm/Group | Treatment Group | Placebo Group
Number analyzed (Participants) | 19 | 19
units on a scale
  MDS-UPDRS 1.3 Depressed Mood | 0.11 [-0.17 to 0.38] | 0.16 [-0.08 to 0.40]
  MDS-UPDRS 1.4 Anxious Mood | -0.16 [-0.53 to 0.21] | 0.21 [-0.05 to 0.47]
  MDS-UPDRS 1.7 Nighttime sleep problems | 0.05 [-0.47 to 0.57] | 1.79 [1.15 to 2.42]

4. Secondary Outcome: Changes in Non-motor Symptoms of PD
Description: Non Motor Symptoms Scale (NMSS) Minimum: 0, maximum: 360, higher score values indicate a worse outcome.
Time Frame: from baseline to 4 weeks + 2 days
Measure: Mean (90% Confidence Interval); unit: score on a scale
Arm/Group | Treatment Group | Placebo Group
Number analyzed (Participants) | 19 | 19
score on a scale | 4.05 [-0.65 to 8.75] | 11.00 [4.68 to 17.32]

5. Secondary Outcome: Changes in Non-motor Symptoms of PD
Description: Hospital anxiety and depression scale (HAD-S) Minimum: 0, maximum: 42, higher score values indicate a worse outcome.
Time Frame: from baseline to 4 weeks + 2 days
Measure: Mean (90% Confidence Interval); unit: units on a scale
Arm/Group | Treatment Group | Placebo Group
Number analyzed (Participants) | 19 | 19
units on a scale
  Hospital anxiety and depression scale - Anxiety | 0.26 [-0.87 to 1.40] | 0.05 [-1.09 to 1.19]
  Hospital anxiety and depression scale - Depression | 0.32 [-1.11 to 1.74] | 0.16 [-0.71 to 1.03]

6. Secondary Outcome: Changes in Non-motor Symptoms of PD
Description: Epworth Sleepiness Scale (ESS) Minimum: 0, maximum: 24, higher score values indicate a worse outcome.
Time Frame: from baseline to 4 weeks + 2 days
Measure: Mean (90% Confidence Interval); unit: units on a scale
Arm/Group | Treatment Group | Placebo Group
Number analyzed (Participants) | 19 | 19
units on a scale | -0.74 [-1.87 to 0.40] | -0.79 [-1.85 to 0.27]

7. Secondary Outcome: Changes in Non-motor Symptoms of PD
Description: Fatigue Severity Scale (FSS) Minimum: 9, maximum: 63, higher score values indicate a worse outcome.
Time Frame: from baseline to 4 weeks + 2 days
Measure: Mean (90% Confidence Interval); unit: units on a scale
Arm/Group | Treatment Group | Placebo Group
Number analyzed (Participants) | 19 | 19
units on a scale | -4.00 [-9.77 to 1.77] | 0.00 [-5.26 to 5.26]

8. Secondary Outcome: Changes in Non-motor Symptoms of PD
Description: King's Parkinson's disease pain scale (KPPS) Minimum: 0, maximum: 168, higher score values indicate a worse outcome.
Time Frame: from baseline to 4 weeks + 2 days
Measure: Mean (90% Confidence Interval); unit: units on a scale
Arm/Group | Treatment Group | Placebo Group
Number analyzed (Participants) | 19 | 19
units on a scale | 1.58 [-2.73 to 5.89] | 2.84 [-5.19 to 10.87]

9. Secondary Outcome: Changes in Non-motor Symptoms of PD
Description: Questionnaire for Impulsive-Compulsive Disorders in Parkinson's Disease-Rating Scale (QUIP-RS) Minimum: 0, maximum: 112, higher score values indicate a worse outcome.
Time Frame: from baseline to 4 weeks + 2 days
Measure: Mean (90% Confidence Interval); unit: units on a scale
Arm/Group | Treatment Group | Placebo Group
Number analyzed (Participants) | 19 | 19
units on a scale | -0.68 [-1.49 to 0.12] | 0.05 [-0.64 to 0.74]

10. Secondary Outcome: Changes in Non-motor Symptoms of PD
Description: Montreal Cognitive Assessment (MoCA) Minimum: 0, maximum: 30, higher score values indicate better outcome.
Time Frame: from baseline to 4 weeks + 2 days
Measure: Mean (90% Confidence Interval); unit: units on a scale
Arm/Group | Treatment Group | Placebo Group
Number analyzed (Participants) | 19 | 19
units on a scale | 0.74 [-0.18 to 1.66] | 0.00 [-0.63 to 0.62]

11. Secondary Outcome: Changes in Non-motor Symptoms of PD
Description: Visual Analog Scale (VAS) of Pain Minimum: 0 mm, maximum: 10 mm, higher score values indicate a worse outcome.
Time Frame: from baseline to 4 weeks + 2 days
Measure: Mean (90% Confidence Interval); unit: millimeters on a scale
Arm/Group | Treatment Group | Placebo Group
Number analyzed (Participants) | 19 | 19
millimeters on a scale | 6.58 [-5.65 to 18.81] | 2.16 [-8.40 to 12.71]

12. Secondary Outcome: Clinical Global Impression - Global Improvement (CGI-I) Scale
Description: Clinical Global Impression - Global Improvement (CGI-I) scale Minimum: 1, maximum: 7, higher score values indicate a worse outcome.
Time Frame: Values of the Termination visit (4 weeks + 2 days from baseline)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Group | Placebo Group
Number analyzed (Participants) | 19 | 19
units on a scale | 4.95 (0.71) | 4.42 (0.61)

13. Secondary Outcome: Incidence of AEs and Number of Withdrawals in PD Patients Taking Nabilone.
Description: Safety and tolerability will be evaluated with reference to the following:
  Number of subjects (%) who discontinue the study Number of subjects (%) who discontinue the study due to AE Adverse Events (AE): total number of patients with all adverse events is reported (no reporting threshold)
Time Frame: from baseline to 4 weeks + 2 days
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group | Placebo Group
Number analyzed (Participants) | 19 | 19
Participants
  Number of subjects who discontinue the study | 0 | 0
  Number of subjects who discontinue due to AEs | 0 | 0
  Total number of patients with Adverse Events | 6 | 8

14. Secondary Outcome: Suicidality in PD Patients Taking Nabilone.
Description: Assessment of aggregated data (suicidality present / no suicidality) of the Columbia-Suicide Severity Rating Scale (C-SSRS). The scale consists of questions for suicidality that can be answered with either "yes" or "no". The answer "no" indicates no wish to be dead, no suicidal ideations, or suicidal attempts.
  No minimum or maximum score values can be provided. The values provided represent the number of patients with (new) suicidality.
Time Frame: from baseline to 4 weeks + 2 days
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group | Placebo Group
Number analyzed (Participants) | 19 | 19
Participants | 0 | 0

15. Secondary Outcome: Change in Hallucinations in PD Patients Taking Nabilone
Description: Number of patients with changes in the points of the Hallucination item (1.2) of the Movement Disorders Society - Unified Parkinson´s Disease Rating Scale (MDS-UPDRS).
Time Frame: from baseline to 4 weeks + 2 days
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group | Placebo Group
Number analyzed (Participants) | 19 | 19
Participants | 0 | 0

16. Secondary Outcome: Orthostatic Hypotension in PD Patients Taking Nabilone
Description: Changes in points of the Orthostatic hypotension (OH) item (1.12) of Movement Disorders Society - Unified Parkinson´s Disease Rating Scale (MDS-UPDRS), minimum of 0, maximum of 4 points, higher score values representing a worse outcome.
Time Frame: from baseline to week 4 + 2 days
Measure: Mean (90% Confidence Interval); unit: units on a scale
Arm/Group | Treatment Group | Placebo Group
Number analyzed (Participants) | 19 | 19
units on a scale | 0.21 [-0.13 to 0.55] | -0.26 [-0.65 to 0.13]

17. Secondary Outcome: Day-time Sleepiness in PD Patients Taking Nabilone: MDS-UPDRS
Description: Changes in points of the Day-time sleepiness item (1.8) of Movement Disorders Society - Unified Parkinson´s Disease Rating Scale (MDS-UPDRS) , minimum of 0, maximum of 4 points, higher score values representing a worse outcome
Time Frame: from baseline to week 4 + 2 days
Measure: Mean (90% Confidence Interval); unit: units on a scale
Arm/Group | Treatment Group | Placebo Group
Number analyzed (Participants) | 19 | 19
units on a scale | 0.26 [-0.01 to 0.53] | 0.11 [-0.21 to 0.42]

18. Secondary Outcome: Subject Incompliance in PD Patients Taking Nabilone
Description: subject incompliance as per drug accountability.
Time Frame: from baseline to week 4 + 2 days
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group | Placebo Group
Number analyzed (Participants) | 19 | 19
Participants | 0 | 0

19. Secondary Outcome: Weight (kg) in PD Patients Taking Nabilone.
Description: changes in weight (kg)
Time Frame: from baseline to week 4 + 2 days
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Treatment Group | Placebo Group
Number analyzed (Participants) | 19 | 19
kg | -0.70 (2.33) | -0.52 (2.37)

20. Secondary Outcome: Changes in Temperature (Degree Celsius) in PD Patients Taking Nabilone.
Description: changes in temperature (degree Celsius)
Time Frame: from baseline to week 4 + 2 days
Measure: Mean (Standard Deviation); unit: degree Celsius
Arm/Group | Treatment Group | Placebo Group
Number analyzed (Participants) | 19 | 19
degree Celsius | 0.17 (0.56) | 0.35 (0.48)

21. Secondary Outcome: Changes in Supine and Standing Blood Pressure Measurements (mmHg) in PD Patients Taking Nabilone.
Description: changes in supine and standing blood pressure measurements (mmHg)
  Row titles:
  1. Mean Change of systolic blood pressure readings (SBP) from supine to standing position for 3 min at the baseline visit
  2. Mean Change of systolic blood pressure readings (SBP) from supine to standing position for 3 min at the week 4 - visit
  3. Mean Change of diastolic blood pressure readings (DBP) from supine to standing position for 3 min at the baseline visit
  4. Mean Change of diastolic blood pressure readings (DBP) from supine to standing position for 3 min at the week 4 - visit
Time Frame: values from baseline and week 4 + 2 days
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Treatment Group | Placebo Group
Number analyzed (Participants) | 19 | 19
mmHg
  Baseline: Change supine - 3 min standing, SBP | 1.47 (13.88) | -4.05 (11.53)
  week4: Change supine - 3 min standing, SBP | -1.84 (10.68) | -2.95 (17.96)
  Baseline: Change supine - 3 min standing, DBP | 3.79 (5.84) | 3.16 (6.07)
  week4: Change supine - 3 min standing, DBP | 4.11 (5.95) | -0.79 (7.90)

22. Secondary Outcome: Changes in Quality of Life of PD
Description: Parkinson´s Disease Questionnaire - 39 (PDQ-39) Minimum: 0, maximum: 156, higher score values indicate a worse outcome. Values were standardized = PDQ-39 Summary Index (SI, the score of each subdomain was divided by the number of questions of that domain and then multiplied by hundred, the sum score is the sum of the results of all 8 domains)
Time Frame: from baseline to week 4 + 2 days
Population: PDQ-39 SI values reported
Measure: Mean (90% Confidence Interval); unit: units on a scale
Arm/Group | Treatment Group | Placebo Group
Number analyzed (Participants) | 19 | 19
units on a scale | -0.49 [-3.04 to 2.05] | -0.47 [-3.21 to 2.28]

23. Other Pre Specified Outcome: The Exploratory Objective of This Study Will be an Eye-tracking Evaluation in PD Patients Taking Nabilone or Placebo.
Description: Change of the reaction time (seconds) between the Screening visit (Part 1) and the Termination visit (Part 2) as measured by the Eye-tracking examination.
Time Frame: Maximum of 104 days
Reporting Status: Not Posted

24. Other Pre Specified Outcome: The Exploratory Objective of This Study Will be an Eye-tracking Evaluation in PD Patients Taking Nabilone or Placebo.
Description: Change of attention span and ability to concentrate (error rate, correct trials) between the Screening visit (Part 1) and the Termination visit (Part 2) as measured by the Eye-tracking examination.
Time Frame: Maximum of 104 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Each patient was assessed from first intake of study drug to study discontinuation.
Description: definitions do not differ
Groups:
- Treatment Group (Open-label Phase); Treatment Group (Double-blind Phase): Nabilone 0.25 mg
  Nabilone 0.25 mg: capsules, 0.25 mg up to 2 mg of nabilone taken orally on a daily basis
- Placebo Group (Double-blind Phase): Placebo (corn starch)
  Placebo: capsule, corn starch, daily basis
Arm/Group | Treatment Group (Open-label Phase) | Treatment Group (Double-blind Phase) | Placebo Group (Double-blind Phase)
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 30/47 | 4/19 | 9/19
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group (Open-label Phase) (N=47) | Treatment Group (Double-blind Phase) (N=19) | Placebo Group (Double-blind Phase) (N=19)
Insomnia (Nervous system disorders) | 0 (0) | 2 (2) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 4 (5) | 0 (0) | 3 (3)
Pain (including worsening) (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) | 2 (2)
Fall (including recurrent falls) (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2)
Fatigue (Nervous system disorders) | 13 (17) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 9 (9) | 0 (0) | 0 (0)
Dry mouth (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0) | 0 (0)
Daytime sleepiness (Nervous system disorders) | 4 (5) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
negative expectations might impact results (due to withdrawal design), sample size of 38 patients (double-blind phase), all caucasian patients

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-08): https://cdn.clinicaltrials.gov/large-docs/96/NCT03769896/Prot_SAP_000.pdf